CLINICAL TRIAL: NCT04135911
Title: A Prospective Study on The"Management of Hypertension in Young and Middle-aged Subjects in Enterprises Setting"
Acronym: PROMISE
Status: Suspended | Type: Observational
Why Stopped: The study was suspended due to limited funding and the COVID-19 pandemic.
Sponsor: Yan Li (Other)
Responsible Party: Sponsor-Investigator, Yan Li, Professor of Cardiovascular Medicine, Shanghai Institute of Hypertension
Organization: Shanghai Institute of Hypertension (Other)
Other Study IDs: PROMISE20190831
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Hypertension; Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In recent years, with the investment from government in the health management of the elderly, community management of hypertension in the elderly has made great progress in management rate and standardized management, but the management of young and middle-aged patients with hypertension is still blank.

Workplace pressure measurement may be more suitable for most of the young and middle-aged patients to find high blood pressure and monitor blood pressure changes in time.

However, there is not much research on workplace pressure measurement. Whether blood pressure measurement in the workplace can reduce the white coat effect, and how it relates to home blood pressure and ambulatory blood pressure is still unclear.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female sex, aged 18-65 years
2. Three different daytime workplace blood pressure measurements meet the limits: systolic blood pressure ≥ 120 mmHg, or diastolic blood pressure ≥80 mmHg
3. Hypertensive patients who are taking antihypertensive drugs
4. Willing to provide information about disease history and lifestyle
5. Willing to receive follow-up for up to 2-3 years
6. Sign the informed consent

Exclusion Criteria:

1. Having the onset of cardiovascular and cerebrovascular diseases such as stroke, myocardial infarction or heart failure within 6 months
2. Having a history of atrial fibrillation or frequent arrhythmia
3. Complicating other diseases that are not suitable for the trial, such as thyroid disease with active medication, acute infectious diseases, chronic mental illness, and tumors
4. The subject is participating in other clinical studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients measuring blood pressure at the workplace with normal high blood pressure or hypertensive patients.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic classification in hypertension | 2 years
  Differences in diagnostic classification between workplace blood pressure and daytime ambulatory blood pressure in the classification of hypertension (masked hypertension or white coat hypertension)

SECONDARY OUTCOMES:
Change in different blood pressure measurement | 2 years
  Differences in workplace blood pressure, daytime ambulatory blood pressure, home blood pressure and 24-hour ambulatory blood pressure
The distribution of heart rate in young and middle-aged subjects | 2 years
  The distribution of heart rate in young and middle-aged subjects who were diagnosed with hypertension
Progression of target organ damage | 2 years
  Differences in the progression of target organ damage between controlled or uncontrolled subjects or between subjects with fast and slow heart rate
The development of with-coat hypertension | 2 years
  The development of white-coat hypertension as persistent hypertension and other types of hypertension or normal blood pressure and changes in target organ damage
The proportion of masked hypertension in patients with normal high blood pressure | 2 years
  The proportion of masked hypertension in patients with normal high blood pressure and the change in outcome after treatment intervention and changes in target organ damage

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China